CLINICAL TRIAL: NCT04771611
Title: COVFIS-HOME: A Phase 2 Placebo-Controlled Pilot Study in COVID-19 of Fisetin to Alleviate Dysfunction and Decrease Complications in At-Risk Outpatients
Brief Title: COVFIS-HOME: COVID-19 Pilot Study of Fisetin to Alleviate Dysfunction and Decrease Complications
Acronym: COVFIS-HOME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James L. Kirkland, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, James L. Kirkland, MD, PhD, Co-Principal Investigator and Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-009705
Record Dates: First submitted 2021-02-24; First posted 2021-02-25 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Covid19; Coronavirus Infection
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Subjects will receive treatment drug Fisetin
  Interventions: Drug: Fisetin
- Placebo (Placebo Comparator): Subjects will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin — ~20mg/kg /day oral for four days (days 0,1 and days 8,9)
  Other Names: 3,3',4',7-tetrahydroxyflavone
  Arms: Treatment Group
Drug: Placebo — Looks exactly like the study drug, but it contains no active ingredient . Oral for four days (days 0,1 and days 8,9)
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether Fisetin, a senolytic drug can assist in the reduction of complications in patients with COVID-19 infection.

DETAILED DESCRIPTION:
To determine whether short-term treatment with Fisetin reduces the rate of death and long term complications related to COVID-19 and to determine the safety of treatment with Fisetin in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 18 years of age, capable and willing to provide informed consent;
* Patient must have received a diagnosis of COVID-19 infection within the last 3 days;
* Outpatient setting (not currently hospitalized);
* Patient must possess at least one of the following high-risk criteria: 60 years or more of age, obesity (BMI ≥ 30 kg/m2), diabetes mellitus, uncontrolled hypertension (systolic blood pressure ≥150 mm Hg), known respiratory disease (including asthma, chronic obstructive pulmonary disease, or present or past smoking), known heart failure, known coronary disease, fever of ≥38.4°C within the last 48 hours, dyspnea at the time of presentation, the combination of high neutrophil count and low lymphocyte count;
* Female patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile, or is of childbearing potential and practicing at least one method of contraception and preferably two complementary forms of contraception including a barrier method (e.g. male or female condoms, spermicides, sponges, foams, jellies, diaphragm, intrauterine device (IUD)) throughout the study and for 30 days after study completion;
* Patient or their caregiver must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

* Patient currently hospitalized or under immediate consideration for hospitalization;
* Patient currently in shock or with hemodynamic instability;
* Patient with severe hepatic disease (as per clinical judgement) and liver enzymes >10x the upper limit of normal;
* Female patient who is pregnant, breast-feeding, or is considering becoming pregnant during the study or for 1 day after the last dose of study medication;
* Patient currently taking Sirolimus, Tacrolimus, or other mTOR inhibitors for other indications (mainly chronic indications represented by organ transplantation or autoimmune diseases);
* On Warfarin therapy;
* Patient with a history of an allergic reaction or significant sensitivity to Fisetin;
* Patient undergoing chemotherapy for cancer;
* Patient is considered by the investigator, for any reason, to be an unsuitable study candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avni Y. Joshi, MD, MS, Principal Investigator — Mayo Clinic; James L Kirkland, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Subjects who received treatment drug Fisetin
  Fisetin: ~20mg/kg /day oral for four days (days 0,1 and days 8,9)
- Placebo: Subjects who received placebo
  Placebo: Looks exactly like the study drug, but it contains no active ingredient. Oral for four days (days 0,1 and days 8,9)
Period: Overall Study
Arm/Group | Treatment Group | Placebo
Started | 29 | 26
Completed | 29 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Placebo | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (15.4) | 58.7 (12.9) | 58.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 26 | 54
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 26 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 26 | 55

OUTCOME MEASURES:

1. Primary Outcome: World Health Organization (WHO) Ordinal Scale Score
Description: The number of subjects who scored as No limitations (Score 0-1) and Ambulatory, limitations (score 2-8) on the WHO Ordinal Scale score. The 9 points of the WHO ordinal clinical severity scale are as follows: 0: no clinical or virological evidence of infection; 1: ambulatory, no activity limitation; 2: ambulatory, activity limitation; 3: hospitalized, no oxygen therapy; 4: hospitalized, oxygen mask or nasal prongs; 5: hospitalized, noninvasive mechanical ventilation (NIMV) or high-flow nasal cannula (HFNC); 6: hospitalized, intubation and invasive mechanical ventilation (IMV); 7: hospitalized, IMV + additional support such as pressors or extracardiac membranous oxygenation (ECMO); 8: death. Total scores range from 0-8. Lower scales indicate less limitations, higher scores indicate more limitations.
Time Frame: 60 days
Population: Two subjects in each arm did not return for the 60-day evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 27 | 24
Participants
  No limitations (Score 0-1) | 26 | 22
  Ambulatory, limitations (score 2-8) | 1 | 2

2. Secondary Outcome: Serious Adverse Events
Description: The number of serious adverse events reported
Time Frame: 60 days
Measure: Number; unit: number of serious adverse events
Arm/Group | Treatment Group | Placebo
Number analyzed (Participants) | 29 | 26
number of serious adverse events | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 60 days.
Arm/Group | Treatment Group | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/29 | 2/26
Other Adverse Events (participants affected / at risk) | 17/29 | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=29) | Placebo (N=26)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Robotic assisted total arthroplasty (right) (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=29) | Placebo (N=26)
Change in stool color (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Infectious Rash (Infections and infestations) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Worsening Headache (Nervous system disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Non cardia chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Systolic murmur (Cardiac disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
ear pain, left (Ear and labyrinth disorders) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
watering eyes (epiphora) (Eye disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
edema, hand, bilateral (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 1 (1)
flu like symptoms (General disorders) | 1 (1) | 1 (1)
Allergy Unspecified (Immune system disorders) | 0 (0) | 1 (1)
Lyme's Disease (Immune system disorders) | 0 (0) | 1 (1)
Vitamin D Deficiency (Immune system disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1)
bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
fatigue (Infections and infestations) | 1 (1) | 0 (0)
pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infections (UTI) (Infections and infestations) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
polyp colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
acute frontal lobe stroke (Nervous system disorders) | 0 (0) | 1 (1)
ageusia (Nervous system disorders) | 1 (1) | 0 (0)
amnesia (Nervous system disorders) | 1 (1) | 0 (0)
migraine (Nervous system disorders) | 1 (1) | 0 (0)
worsening Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
anxiety attack (Psychiatric disorders) | 0 (0) | 1 (1)
Colic Renal (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis Calcium Oxalate (Renal and urinary disorders) | 1 (1) | 0 (0)
bacterial vaginosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
asthma with exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
change in smell (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
thrush (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
arthoplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
right shoulder arthroscopy, rotator cuff, repair (Surgical and medical procedures) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT04771611/Prot_SAP_000.pdf